CLINICAL TRIAL: NCT04985513
Title: Electrical Impedance Tomography Based Regional Lung Ventilation Evaluation According to Ventilation Strategy During Cardiopulmonary Bypass in Minimally Invasive Cardiac Surgery
Brief Title: EIT Based Regional Lung Ventilation in Minimally Invasive Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Hyung Gon Je, Associate professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 05-2021-156
Record Dates: First submitted 2021-07-16; First posted 2021-08-02 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Patients Who Underwent CPB for MICS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (No Intervention): Stopping ventilation during cardiopulmonary bypass
- Group V (Active Comparator): Ventilation was performed using an inhaled oxygen fraction of 20% and a tidal volume of 5ml/kg at the time of cardiopulmonary bypass.
  Interventions: Procedure: Ventilation during cardiopulmonary bypass

INTERVENTIONS:
Procedure: Ventilation during cardiopulmonary bypass — Ventilation was performed using an inhaled oxygen fraction of 20% and a tidal volume of 5ml/kg at the time of cardiopulmonary bypass.
  Arms: Group V

SUMMARY:
Electrical impedance tomography (EIT) is a non-invasive, radiation-free imaging technique that measures local pulmonary ventilation and ventilation distribution through potential changes on the skin surface of the chest wall during the respiratory cycle. Recently, a global inhomogeneity (GI) index has been proposed and used to quantify the distribution of tidal volume in the lungs. Currently, there are research results showing that ventilation improves postoperative oxygenation and gas exchange when ventilation is applied during CPB, but the evidence for long-term prognosis is lacking. In this study, researchers performed electrical impedance tomography in the intensive care unit immediately after surgery on patients who had undergone endotracheal tube extubation in the operating room immediately after completing minimally invasive cardiac surgery by collapsing the right lung through right minimal thoracotomy. The purpose of this study is to measure local pulmonary ventilation and ventilation distribution using this method and to find the optimal left lung ventilation method during minimally invasive cardiac surgery based on this. Identifying the difference in postoperative pulmonary ventilation disorders and functional regional ventilation according to the pulmonary ventilation strategy at the time of CPB in minimally invasive cardiac surgery can help predict the risk of pulmonary complications and improve the prognosis of patients after surgery.

DETAILED DESCRIPTION:
Minimally invasive cardiac surgery (MICS) is a safe and effective surgical method that reduces bleeding, number of reoperations, postoperative pain, and length of stay in the ICU, and promotes faster recovery compared to conventional open thoracic cardiac surgery. In general, since cardiopulmonary bypass (CPB) is used during minimally invasive cardiac surgery using right thoracotomy, both lungs can be maintained in a lung rest state. Except for 2-3 ventilations when releasing the aortic forceps during surgery, there is no ventilation at all during CPB, and both lung ventilation starts when CPB is stopped. In order to secure the surgical field of view during surgery, most anesthetists do not ventilate the right lung and maintain a collapsed state. Even during CPB, ventilation can be performed without affecting the field of vision at the surgical site. However, to date, it is not well known about the proper ventilation method for the left lung during cardiac surgery using CPB.

Pulmonary complications are major postoperative complications of minimally invasive cardiac surgery and are factors that increase postoperative pulmonary complications, such as age, preoperative lung disease, and duration of CPB, which are well-known. Failure to ventilate the entire lung field at the time of CPB may cause atelectrauma, and even if normal ventilation is performed after CPB, and shearing force from repeated collapse and expansion of the atelectasis area may occur. In addition, such atelectasis can lead to not only ventilation disorders, ventilation/perfusion imbalances, but also postoperative pneumonia and poor prognosis. In particular, since right thoracotomy is mainly performed in minimally invasive cardiac surgery, the right lung collapses through one lung ventilation from the start of the operation to the access to the surgical site or at the end of the operation to check for bleeding at the surgical site. Therefore, one lung ventilation may be required even after weaning from the CPB, which may increase the risk of atelectasis in the operated side. Depending on the ventilation of the left lung during surgery and the tidal volume (TV), it may affect postoperative atelectasis and may cause functional ventilation. This can lead to the occurrence of respiratory complications such as pneumonia after surgery, resulting in poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 18 years of age
2. Patients who underwent one lung ventilation using a bronchial blocker for minimally invasive cardiac surgery
3. If there is no atelectasis on chest X-ray or chest computed tomography performed before surgery

Exclusion Criteria:

1. If there is evidence of atelectasis, pneumonia, or lung disease that can reduce lung volume in a chest X-ray examination or chest computed tomography performed before surgery
2. Patients scheduled for sternotomy
3. If there is a skin disease in the chest that requires EIT measurement
4. If there is a plan to transfer to the intensive care unit while maintaining the endotracheal tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
postoperative pulmonary ventilation disorders | after ICU transferring (up to 1hour)
  Confirmation of postoperative pulmonary ventilation disorders according to the lung ventilation strategy at the time of cardiopulmonary bypass in minimally invasive cardiac surgery

SECONDARY OUTCOMES:
incidence of postoperative pulmonary complications | during ICU hospitalization (up to 7 days)
  the difference in the incidence of postoperative pulmonary complications according to the pulmonary ventilation strategy at the time of cardiopulmonary bypass in minimally invasive cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Gon Je, Principal Investigator — School of Medicone, Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

REFERENCES:
- [Derived] Yeo HJ, Kim HY, Je HG, Kim HJ, Park S, Yoon JP, Ju MH, Lim MH, Lee CH. Electrical impedance tomography-based evaluation of regional lung ventilation according to ventilation strategy during cardiopulmonary bypass in minimally invasive cardiac surgery: a prospective randomized controlled trial. J Thorac Dis. 2025 Jun 30;17(6):3912-3923. doi: 10.21037/jtd-24-1877. Epub 2025 Jun 23. PMID 40688333